CLINICAL TRIAL: NCT05748522
Title: Functional Movement Analysis (FMS) of Diaphragmatic Breathing-Immediate Effect on Shoulder Mobility- Randomized Controlled, Single-Blind Study
Brief Title: Functional Movement Analysis (FMS) of Diaphragmatic Breathing-Immediate Effect on Shoulder Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-240
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Pain; Diaphragm Issues
Keywords: Diaphragmatic Breathing; Functional Movement Analysis (FMS); Shoulder Mobility
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder Mobility (Other): It is one of the seven functional movements studied in FMS. This test requires the participant to simultaneously hold one hand behind the back (internal rotation) and the other hand behind the head (external rotation) with the fisted hands, and bring the hands as close to each other as possible in the back area. The distance measurement in cm is taken with a tape measure between 3 fingers of both hands. This type of reach test has been described as a tool for measuring glenohumeral joint (GH) mobility through functional shoulder movements.
  Interventions: Procedure: Diaphragmatic Breathing
- Diaphragmatic Breathing (Experimental): The participant lies on his back. He places his hands horizontally on the lowest part of the ribs. While inhaling, he is asked to inflate his stomach towards the bottom of his hands. It is taught that during breathing, the abdomen should swell rather than the rib cage, and the ribs should open outwards. Breath is taken through the nose, blown slowly through the mouth.
  Interventions: Other: Shoulder Mobility

INTERVENTIONS:
Other: Shoulder Mobility — t is one of the seven functional movements studied in FMS. This test requires the participant to simultaneously hold one hand behind the back (internal rotation) and the other hand behind the head (external rotation) with the fisted hands, and bring the hands as close to each other as possible in the back area. The distance measurement in cm is taken with a tape measure between 3 fingers of both hands.
  Arms: Diaphragmatic Breathing
Procedure: Diaphragmatic Breathing — The participant will lie on his back in a comfortable position, diaphragmatic breathing will be taught first in the application group and he will be asked to do diaphragmatic breathing for 90 seconds. At the end of this period, the participant will be referred back to the evaluator physiotherapist, and the physiotherapist will evaluate the shoulder mobility again without knowing which group the participant is in.
  In the participant control group, shoulder mobility will be evaluated and the practitioner will be asked to stay in a comfortable position on his back for 90 seconds next to the physiotherapist. At the end of the period, shoulder mobility will be evaluated again by the assessing physiotherapist.
  Arms: Shoulder Mobility

SUMMARY:
The diaphragm is defined as a thin, smooth muscle that separates the thoracic and abdominal cavities. The shoulder and diaphragm muscle have a clear relationship through innervation and myofascial tissue connection. Fascia is often neglected medically, rehabilitatively, or performance as the underlying cause of problems. Bones, organs, and muscles appear to float in the fascial web, a continuous three-dimensional system of connective tissue. Plastic and viscoelastic properties, which can change tension and shape under the influence of manual techniques and movement retraining, ensure that the structural changes are reversible. Functional Movement Analysis (FMS) is a screening system that aims to predict the risk of injury and functional deficiencies. FMS consists of 7 basic motion component tests. It is scored on a scale of zero to three and creates a composite score whose sum ranges from 0 to 21 points. One of the 7 motion models evaluated is shoulder mobility. According to the results of this study, people who perform activities that require shoulder mobility will be guided as to whether the use of diaphragmatic breathing will be effective for preparation, rehabilitation or performance improvement. The aim of the study was to observe whether shoulder mobility increased in healthy individuals taught diaphragm breathing compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Individuals between the ages of 18-30

Exclusion Criteria:

* Have a musculoskeletal injury/operation involving the shoulder area in the last 6 months
* Using drugs that can affect the respiratory system
* Have received aerobic exercise training in the last 6 weeks

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Shoulder Mobility Measurement | 4 weeks
  It is one of the seven functional movements studied in FMS. This test requires the participant to simultaneously hold one hand behind the back (internal rotation) and the other hand behind the head (external rotation) with the fisted hands, and bring the hands as close to each other as possible in the back area. The distance measurement in cm is taken with a tape measure between 3 fingers of both hands.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided